CLINICAL TRIAL: NCT03617211
Title: A Multi-center Study: The Follow-up of Complications for Women Having Pelvic Reconstruction Surgery With Mesh/Native Tissue(Part II).
Brief Title: The Follow-up of Mesh/Native Tissue Complications Study(Part II)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University People's Hospital (Other); Qilu Hospital of Shandong University (Other); Obstetrics & Gynecology Hospital of Fudan University，Shanghai Red House Obstetrics & Gynecology Hospital (Unknown); Peking University Third Hospital (Other); First Hospitals affiliated to the China PLA General Hospital (Other Government); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Tongji Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Wuxi Obsetrics & Gynecology Hospital (Unknown); Fuzhou General Hospital (Other); The First Affiliated Hospital of Jinan Hospital (Unknown); Women's Hospital School Of Medicine Zhejiang University (Other); Renmin Hospital of Wuhan University (Other); The Third Hospital Affiliated Zhengzhou University (Unknown); Shengjing Hospital (Other); General Hospital of Ningxia Medical University (Other); The Second Hospital of Hebei Medical University (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Yantai Yuhuangding Hospital，Medical College, Qingdao University (Unknown); Southwest Hospital, China (Other); West China Second University Hospital (Other); Jiangxi Maternal and Child Health Hospital (Other); Chongqing Medical University (Other); Shanxi Coal Central Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: JS-1566-2
Record Dates: First submitted 2018-07-12; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-06

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic reconstructive surgery; mesh; native tissue; tape; complications; Category-time-site (CTS) coding
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study the incidence and distribution of complications after different pelvic reconstruction surgeries (mesh/native tissue) in multi-centers. The investigators aimed to report and summarize the postoperative complications diagnosed in the prior 1 year, 3 years and 5 years respectively, according to the International Urogynecological AssociationInternational Continence Society(IUGA-ICS) Complication Classification Coding(Category-Time-Site coding system) .

DETAILED DESCRIPTION:
Patients are inferred to 27 tertiary hospitals with the complaint of de novo complications after pelvic reconstructive surgeries using mesh, tape and native tissue between June 2018 and June 2023. The subjects include patients who accept treatment not only at 27 participating hospitals but also from other hospital. And the date of surgeries carried is not restricted in the study period.

This is a study of real world. The researchers focus to investigate the incidence of complications in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients are inferred to the clinic with the complaint of de novo complications after pelvic reconstructive surgeries with mesh,tape or native tissue.
* 2) Pelvic reconstructive surgeries include but not limited to open/laparoscopic sacrocolpopexy (Y-shape tape/self-cut synthesized mesh), anterior, apical, posterior or total pelvic reconstruction with trans-vaginal mesh(commercial mesh kits or self-cut synthesized mesh), repair using native tissue(sacrospinous ligament fixation, high uterosacral ligament suspension, ischial spinous fascia fixation, the Lefort operation) and as well as anti-urinary incontinence surgeries(tension-free vaginal tape).
* 3) Both primary and repeated pelvic surgery are included.

Exclusion Criteria:

* If the same patient who developed complications after pelvic floor reconstructive surgeries has been diagnosed and reported in 27 participating hospitals, and again treated for "the same code complication in other 26 hospitals, she will be ruled out.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are inferred to 27 tertiary hospitals with the complaint of de novo complications after pelvic reconstructive surgeries using mesh, tape and native tissue between June 2018 and June 2023. The subjects include patients who accept treatment not only at our participating hospitals but also from other hospital.And the date of surgeries carried is not restricted during the study period.
Sampling Method: Probability Sample
Enrollment: 1530 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The frequency and ratio of different postoperative complications | 1-year;3-year;5-year
  Calculate the frequency(reported in number of cases) and ratio(reported in percentage, %) of different complications reported from 27 tertiary hospitals in the past year or 3 years or 5 years, respectively.The complications occurred after pelvic reconstructive surgeries, especially mesh/native tissue related,are classified by IUGA-ICS CTS(category-time-site)coding system.

SECONDARY OUTCOMES:
The distribution of complications after each kind of pelvic reconstructive surgery | 1-year;3-year;5-year
  For each kind of surgery,the distribution of different postoperative complications, classified by the IUGA-ICS coding system, is expressed in frequency (reported in number of cases) and ratio(reported in percentage, %).
The percentage of various pelvic reconstructive surgeries under the same complication classification coding. | 1-year;3-year;5-year
  Analyze and calculate the percentage of different surgical method when they present the complication with the same IUGA-ICS coding.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, MD, Principal Investigator — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences
Locations (5):
- China (5):
  - First Affiliated Hospital of PLA General Hospital (304), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Wuxi Obstetrics & Gynecology Hospital, Wuxi, Jiangsu
  - Obstetrics & Gynecology Hospital of Fudan University，Shanghai Red House Obstetrics & Gynecology Hospital, Shanghai, Shanghai Municipality